CLINICAL TRIAL: NCT06542159
Title: Elimination of PTV Margins Based on Online Adaptive Stereotactic Radiotherapy for Early-stage Non-small Cell Lung Cancer or Pulmonary Oligometastases: a Prospective, Randomized, Controlled Phase II Study
Brief Title: Elimination of PTV Margins Based on Online Adaptive Stereotactic Radiotherapy for Early-stage Non-small Cell Lung Cancer or Pulmonary Oligometastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-10116
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Adaptive Radiotherapy; Stereotactic Body Radiotherapy; Non-small Cell Lung Cancer; Lung Oligometastases; Toxicity
Keywords: Online adaptive radiotherapy; Stereotactic body radiotherapy; Non-small Cell Lung Cancer; Lung oligometastases; Toxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group (Experimental): Patients in the study group will receive online adaptive stereotactic body radiotherapy (without PTV expansion margin). The total dose will be 45-50Gy/3-4 fractions, administered once daily. Both FBCT and 4DCT will be acquired before initiating treatment at each fraction.
  Interventions: Radiation: Online adaptive SBRT
- The control group (Active Comparator): Patients in the control group will receive conventional standard stereotactic body radiotherapy. The total dose will be 45-50Gy/3-4 fractions, administered once daily. CBCT will be acquired before initiating treatment at each fraction.
  Interventions: Radiation: Conventional SBRT

INTERVENTIONS:
Radiation: Online adaptive SBRT — Online adaptive SBRT (without PTV expansion margin). The total dose will be 45-50Gy/3-4 fractions, administered once daily. FBCT and 4DCT will be acquired.
  Arms: The study group
Radiation: Conventional SBRT — SBRT with PTV expansion. The total dose will be 45-50Gy/3-4 fractions, administered once daily. CBCT will be acquired.
  Arms: The control group

SUMMARY:
This study aims to explore the safety and efficacy of eliminating the PTV (planning target volume) margins based on online adaptive stereotactic radiotherapy for patients with early-stage non-small cell lung cancer (NSCLC) or pulmonary oligometastases.

DETAILED DESCRIPTION:
This study aims to explore the safety and efficacy of eliminating the PTV expansion margin based on online adaptive stereotactic body radiotherapy (SBRT) for early-stage non-small cell lung cancer (NSCLC) or pulmonary oligometastases. In this study, patients will be stratified according to whether they have primary early-stage NSCLC, then randomly assigned in a 1:1 ratio to the study group or the control group. Patients in the study group will receive online adaptive SBRT (without PTV expansion margin), while patients in the control group will receive conventional standard SBRT. After the completion of treatment, patients will be followed up regularly to assess safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or PET-CT confirmed untreated early-stage non-small cell lung cancer (T1-2N0M0) that is inoperable or where the patient is unwilling to undergo surgery, or PET-CT/chest CT confirmed lung oligometastases (number of metastases ≤3, single lesion diameter ≤5cm).
* Age 18 years or older, regardless of gender.
* ECOG performance status score of 0-2.
* Serum hemoglobin ≥ 80 g/L, platelets ≥ 100,000/μL, absolute neutrophil count ≥ 1,500/μL.
* Serum creatinine ≤ 1.25 times the upper normal limit (UNL) or creatinine clearance ≥ 60 ml/min.
* Serum bilirubin ≤ 1.5 times UNL, AST (SGOT) and ALT (SGPT) ≤ 2.5 times UNL, alkaline phosphatase ≤ 5 times UNL.
* FEV1 ≥ 0.5 L.
* Normal CB6 range.
* The patient and their family agree and sign the informed consent form.

Exclusion Criteria:

* Tumors with bronchial invasion are excluded.
* Any other disease or condition that contraindicates radiotherapy (e.g., active infections, within 6 months post-myocardial infarction, symptomatic heart disease including unstable angina, congestive heart failure, or uncontrolled arrhythmias).
* Pregnant or breastfeeding women, women who have not undergone pregnancy testing, and pregnant individuals.
* Individuals with substance abuse issues, chronic alcoholism, or AIDS.
* Individuals with uncontrollable seizures or loss of self-control due to psychiatric disorders.
* Individuals with a history of severe allergies or specific sensitivities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2027-04-21 (Estimated); Study Completion 2028-04-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2 or higher respiratory toxicity | 1 year
  Incidence of grade 2 or higher respiratory toxicity

SECONDARY OUTCOMES:
Objective response rate | 2 months after radiotherapy
  Objective Response Rate (ORR) is defined as the proportion of patients whose tumor size decreases to a pre-specified value and is maintained for a certain period of time during cancer treatment. It includes the number of patients with Complete Response (CR) and Partial Response (PR) as a percentage of the total number of evaluable cases.
Local control rate | 2 year
  The control of the local lesion after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ganti AK, Klein AB, Cotarla I, Seal B, Chou E. Update of Incidence, Prevalence, Survival, and Initial Treatment in Patients With Non-Small Cell Lung Cancer in the US. JAMA Oncol. 2021 Dec 1;7(12):1824-1832. doi: 10.1001/jamaoncol.2021.4932. PMID 34673888
- [Background] Prezzano KM, Ma SJ, Hermann GM, Rivers CI, Gomez-Suescun JA, Singh AK. Stereotactic body radiation therapy for non-small cell lung cancer: A review. World J Clin Oncol. 2019 Jan 10;10(1):14-27. doi: 10.5306/wjco.v10.i1.14. PMID 30627522
- [Background] Sun B, Brooks ED, Komaki RU, Liao Z, Jeter MD, McAleer MF, Allen PK, Balter PA, Welsh JD, O'Reilly MS, Gomez D, Hahn SM, Roth JA, Mehran RJ, Heymach JV, Chang JY. 7-year follow-up after stereotactic ablative radiotherapy for patients with stage I non-small cell lung cancer: Results of a phase 2 clinical trial. Cancer. 2017 Aug 15;123(16):3031-3039. doi: 10.1002/cncr.30693. Epub 2017 Mar 27. PMID 28346656
- [Background] Timmerman RD, Hu C, Michalski JM, Bradley JC, Galvin J, Johnstone DW, Choy H. Long-term Results of Stereotactic Body Radiation Therapy in Medically Inoperable Stage I Non-Small Cell Lung Cancer. JAMA Oncol. 2018 Sep 1;4(9):1287-1288. doi: 10.1001/jamaoncol.2018.1258. PMID 29852036
- [Background] Adebahr S, Collette S, Shash E, Lambrecht M, Le Pechoux C, Faivre-Finn C, De Ruysscher D, Peulen H, Belderbos J, Dziadziuszko R, Fink C, Guckenberger M, Hurkmans C, Nestle U. LungTech, an EORTC Phase II trial of stereotactic body radiotherapy for centrally located lung tumours: a clinical perspective. Br J Radiol. 2015 Jul;88(1051):20150036. doi: 10.1259/bjr.20150036. Epub 2015 Apr 15. PMID 25873481
- [Background] Roach MC, Robinson CG, DeWees TA, Ganachaud J, Przybysz D, Drzymala R, Rehman S, Kashani R, Bradley JD. Stereotactic Body Radiation Therapy for Central Early-Stage NSCLC: Results of a Prospective Phase I/II Trial. J Thorac Oncol. 2018 Nov;13(11):1727-1732. doi: 10.1016/j.jtho.2018.07.017. Epub 2018 Jul 26. PMID 30056162
- [Background] Bezjak A, Paulus R, Gaspar LE, Timmerman RD, Straube WL, Ryan WF, Garces YI, Pu AT, Singh AK, Videtic GM, McGarry RC, Iyengar P, Pantarotto JR, Urbanic JJ, Sun AY, Daly ME, Grills IS, Sperduto P, Normolle DP, Bradley JD, Choy H. Safety and Efficacy of a Five-Fraction Stereotactic Body Radiotherapy Schedule for Centrally Located Non-Small-Cell Lung Cancer: NRG Oncology/RTOG 0813 Trial. J Clin Oncol. 2019 May 20;37(15):1316-1325. doi: 10.1200/JCO.18.00622. Epub 2019 Apr 3. PMID 30943123
- [Background] Haasbeek CJ, Lagerwaard FJ, Slotman BJ, Senan S. Outcomes of stereotactic ablative radiotherapy for centrally located early-stage lung cancer. J Thorac Oncol. 2011 Dec;6(12):2036-43. doi: 10.1097/JTO.0b013e31822e71d8. PMID 21892102
- [Background] Chen H, Laba JM, Zayed S, Boldt RG, Palma DA, Louie AV. Safety and Effectiveness of Stereotactic Ablative Radiotherapy for Ultra-Central Lung Lesions: A Systematic Review. J Thorac Oncol. 2019 Aug;14(8):1332-1342. doi: 10.1016/j.jtho.2019.04.018. Epub 2019 May 7. PMID 31075543
- [Background] Verma V, Shostrom VK, Kumar SS, Zhen W, Hallemeier CL, Braunstein SE, Holland J, Harkenrider MM, S Iskhanian A, Neboori HJ, Jabbour SK, Attia A, Lee P, Alite F, Walker JM, Stahl JM, Wang K, Bingham BS, Hadzitheodorou C, Decker RH, McGarry RC, Simone CB 2nd. Multi-institutional experience of stereotactic body radiotherapy for large (>/=5 centimeters) non-small cell lung tumors. Cancer. 2017 Feb 15;123(4):688-696. doi: 10.1002/cncr.30375. Epub 2016 Oct 14. PMID 27741355
- [Background] Qin Y, Zhang F, Yoo DS, Kelsey CR, Yin FF, Cai J. Adaptive stereotactic body radiation therapy planning for lung cancer. Int J Radiat Oncol Biol Phys. 2013 Sep 1;87(1):209-15. doi: 10.1016/j.ijrobp.2013.05.008. Epub 2013 Jun 19. PMID 23790773
- [Background] Meng Y, Luo W, Xu H, Wang W, Zhou S, Tang X, Li Z, Zhou C, Yang H. Adaptive intensity-modulated radiotherapy with simultaneous integrated boost for stage III non-small cell lung cancer: Is a routine adaptation beneficial? Radiother Oncol. 2021 May;158:118-124. doi: 10.1016/j.radonc.2021.02.019. Epub 2021 Feb 23. PMID 33636232
- [Background] Zhou S, Meng Y, Sun X, Jin Z, Feng W, Yang H. The critical components for effective adaptive radiotherapy in patients with unresectable non-small-cell lung cancer: who, when and how. Future Oncol. 2022 Oct;18(31):3551-3562. doi: 10.2217/fon-2022-0291. Epub 2022 Oct 3. PMID 36189758
- [Background] Snyder J, Smith B, Aubin JS, Shepard A, Hyer D. Simulating an intra-fraction adaptive workflow to enable PTV margin reduction in MRIgART volumetric modulated arc therapy for prostate SBRT. Front Oncol. 2024 Jan 8;13:1325105. doi: 10.3389/fonc.2023.1325105. eCollection 2023. PMID 38260830
- [Background] Dohopolski M, Visak J, Choi B, Meng B, Parsons D, Zhong X, Inam E, Avkshtol V, Moon D, Sher D, Lin MH. In silico evaluation and feasibility of near margin-less head and neck daily adaptive radiotherapy. Radiother Oncol. 2024 Aug;197:110178. doi: 10.1016/j.radonc.2024.110178. Epub 2024 Mar 6. PMID 38453056